CLINICAL TRIAL: NCT04337099
Title: A Single Patient Compassionate Use of MBM-02 (Tempol) for the Treatment of Prostate Cancer
Status: Available | Type: Expanded Access
Sponsor: Matrix Biomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MBI-11-01
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tempol; TEMPOL-H

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: MBM-02 (Tempol) — Study drug will be administered orally using the capsule formulation (200 mg). The study drug will be administered 7 days a week for the entire treatment period.
  Other Names: Tempol; 4-hydroxy-tempo; 4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl

SUMMARY:
A single patient compassionate use clinical trial for the use of MBM-02 (TEMPOL) for the treatment of prostate cancer. The single patient will be exposed to orally administered TEMPOL for up to 12 months at a maximum total daily dose of 800mg.

DETAILED DESCRIPTION:
Localized therapy for prostate cancer is often curative; however, 20% to 30% of patients experience a recurrence. Biochemical recurrence (BCR) occurs in an estimated 50,000 men/year in the U.S and is marked by a rising prostate specific antigen (PSA) after definitive radical prostatectomy and/or radiation therapy for localized disease.

Continuous androgen deprivation therapy (ADT), in which serum testosterone is decreased to a castrate level (less than 50 ng/dL) is a standard treatment in BCR. ADT is associated with significant short term and long term toxicities, including declining quality of life on treatment and increased risk of osteoporosis, diabetes, and cardiovascular disease. MBM-02 is being tested as a novel non-hormonal agent with improved biologic activity and better tolerability for use in biochemically recurrent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical Recurrent Prostate Cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Prostate Oncology Specialists, Marina del Rey, California, United States

REFERENCES:
- See also: Matrix Biomed, Inc. Compassionate Use — http://matrixbiomed.com/compassionate-use/